CLINICAL TRIAL: NCT05825118
Title: Neutrophil-lymphocyte Ratio Versus Lactate-albumin Ratio as a Predictor of Morbidity and Mortality in Patients With Sepsis and Septic Shock
Brief Title: N\L Ratio Versus L\A Ratio as a Predictor of Morbidity and Mortality in Sepsis and Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Walaa Adel Abdelghafar Elbialy, Principal Investigator, Tanta University
Other Study IDs: N\L and L\A in sepsis
Record Dates: First submitted 2023-03-27; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-03

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Diagnostic Test: Neutrophil/Lymphocyte ratio and lactate/ albumin ratio will be measured in all patients. — Blood will be drawn from peripheral vein, arterial or a central catheter for evaluation of whole blood count, serum lactate and serum albumin.

SUMMARY:
The aim of the study is to compare between neutrophil lymphocyte ratio and lactate albumin ratio as a predictor of morbidity and mortality in sepsis and septic shock patients.

DETAILED DESCRIPTION:
Sepsis is a systemic inflammatory response syndrome caused by infection can lead to life threatening multi-organ dysfunction.

Septic shock causes circulatory and metabolic abnormalities, leading to increased mortality in hospitalized patients, especially in intensive care unit (ICU) patients.

Sepsis can affect the function and number of immune cells, including neutrophils, lymphocytes and monocytes.

Neutrophils play crucial roles in the innate cellular immune system. Early higher neutrophil counts correlated with increased sepsis severity.

In sepsis, lymphocytes decrease owing to the apoptosis mediated by innate response.

Reversily, number of neutrophils dramatically increase reflecting degree of inflammation.

The neutrophil-to-lymphocyte ratio (NLR) is a novel inflammatory biomarker that can be obtained through blood routine tests, it is cost- effective and widely available, and it is beneficial to the early recognition of poor prognosis in septic patients.

Albumin is a molecule that is the most abundant protein in plasma. For a variety of physiological mechanisms, albumin has a variety of function, including serving as a major buffer, extracellular antioxidant, immune modulator, antidote and transporter in plasma.

Increased capillary leakage of albumin is one of the features of SIRS. This means that lower albumin levels correlate with severe systemic inflammation and organ failure.

Hypoxia and tissue hypo perfusion seen in sepsis play a key role on the development of multi-organ failure in septic patients.

Lactic acidosis is one of the best indicators of the insufficient perfusion or development of anaerobic metabolism during septic shock.

The inability of liver to metabolize lactate as a result of the deterioration of liver perfusion also increases lactate levels.

The measurement of blood lactate levels used to determine tissue hypoxia is rapid, inexpensive and easy.

Because lactate and albumin levels progress differently as the development of sepsis proceeds, a ratio between the two rather than analyzing lactate and albumin alone may be a new and perhaps better indicator for the patient's prognosis.

ELIGIBILITY:
Inclusion Criteria

* Age from 18 to 60 years old.
* Patients with suspected infection who fulfilled at least two of three quick sepsis - related organ failure assessment (QSOFA) criteria
* Patients with Organ dysfunction can be confirmed by acute change in SOFA score variables >2 points consequent to infection.
* Sepsis with persisting hypotension requiring vasopressors to maintain MAP > 65 mm Hg and having a serum lactate level > 2mmol/L despite adequate volume of resuscitation.

Exclusion criteria

* No informed consent.
* Malignancy and chemotherapy during the previous 90 days.
* History of steroid therapy within 3 months before admission.
* Patients with either established hepatic dysfunction, renal failure, having any disease in which albumin should be supplemented as liver cirrhosis with ascites, nephrotic syndrome and burn.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: All patient of both sex with age between 18-60 years old admitted to SICU suffering from sepsis and septic shock will be enrolled in the study after fulfillment of the following inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Prediction of 28 day mortality. | 28 days
  Prediction of 28 day mortality (patients will be followed by telephone for 28 day after discharge).

SECONDARY OUTCOMES:
Extent of organ dysfunction in patients with sepsis and septic shock assessed by SOFA score | 0 hours, 6 hours, 24 hours of admission to icu
  SOFA score for assessment of organ dysfunction in 0 hours, 6 hours, 24 hours of admission to icu.

CONTACTS AND LOCATIONS:
Overall Officials: Sabry M Ameen, professor, Study Chair — Tanta University; Ahmed A abdelhafez, assist. pro, Study Director — Tanta University; Alaa M Abohagar, lecturer, Principal Investigator — Tanta University
Locations (1):
- Tanta U, Tanta, Egypt

REFERENCES:
- [Background] Fortini A, Faraone A, Meini S, Bettucchi M, Longo B, Valoriani B, Forni S; Italian Federation of Hospital Internists (FADOI) - Sepsis Collaboration Group of the Tuscany Region. Validity of "Sepsis-3" criteria in identifying patients with community-onset sepsis in Internal Medicine wards; a prospective, multicenter study. Eur J Intern Med. 2021 Mar;85:92-97. doi: 10.1016/j.ejim.2020.12.025. Epub 2021 Jan 12. PMID 33451890
- [Background] Gaieski DF, Edwards JM, Kallan MJ, Carr BG. Benchmarking the incidence and mortality of severe sepsis in the United States. Crit Care Med. 2013 May;41(5):1167-74. doi: 10.1097/CCM.0b013e31827c09f8. PMID 23442987
- [Background] Cao C, Yu M, Chai Y. Pathological alteration and therapeutic implications of sepsis-induced immune cell apoptosis. Cell Death Dis. 2019 Oct 14;10(10):782. doi: 10.1038/s41419-019-2015-1. PMID 31611560